CLINICAL TRIAL: NCT06350240
Title: Investigation of the Effects of Textured Insoles and Exercise on Tactile Sense, Balance, Foot Load Distribution and Quality of Life in Children With Joint Hypermobility
Brief Title: Effects of Textured Insoles and Exercise in Children With Joint Hypermobility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Kamile Uzun Akkaya, PhD, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUzunAkkaya
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Child, Only; Joint Laxity; Exercise; Textured Insoles
MeSH Terms: conditions — Joint Instability; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): Exercise group
  Interventions: Behavioral: Exercise
- Intervention group (Experimental): Exercise and use of textured insoles group
  Interventions: Behavioral: Exercise+texture insoles

INTERVENTIONS:
Behavioral: Exercise — An exercise program that can be easily applied at home and in the park, which will support the psychomotor, tactile and proprioceptive-rich sensory development specific to children with joint hypermobility. The family will be instructed to do these exercises for 30 minutes a day for 5 days in total, 2 days a week in the playground and 3 days at home for 6 weeks, and the family will be asked to keep a diary to see whether they do the exercises or not.
  Arms: Control group
Behavioral: Exercise+texture insoles — In addition to exercise, children in this group will have an individual textured insoles made to suit the child's foot. The child will be asked to place textured insoles inside his shoes and use the textured insoles for 6-8 hours.
  Arms: Intervention group

SUMMARY:
Joint hypermobility is the condition that the joints have a greater range of motion than normal and can be observed frequently in children. In children with joint hypermobility, motor problems, tactile and proprioceptive sensory disorders can be observed. It is very important to support children with joint hypermobility with intervention programs that are rich in both motor and sensory aspects. The aim of this project is to create an exercise protocol rich in tactile, proprioceptive senses for children with joint hypermobility and to examine the effects of using textured insoles in addition to exercise on tactile sense, balance, foot load distribution and quality of life in children.

DETAILED DESCRIPTION:
It was planned to include 40 children with joint hypermobility in the project. Children's joint hypermobility will be determined by the Beighton Score. Children will be divided into two groups. Children in both groups will be offered an exercise program consisting of home and park activities that will improve their motor and sensory aspects. Children in the intervention group will be asked to additionally use textured insoles. Before and after the study, children's plantar foot tactile sense, balance, foot load distribution and quality of life will be evaluated. Pre- and post-treatment values and change values in both groups will be compared with each other.

ELIGIBILITY:
Inclusion Criteria:

* Children with a Beighton score of 6 and above
* Being between the ages of 5-18
* Being cooperative in the assessments and treatment
* Having a body mass index between 18.5-24.9

Exclusion Criteria:

* Having had any surgery or trauma in the last 6 months
* Having any neurological, metabolic, rheumatological or chronic disease.
* Having a vestibular system problem
* Being diagnosed with Ehlers-Danlos Syndrome
* Having foot wounds and anomalies that may affect sole sensation
* Having chronic pain.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Tactile sense | Through study completion, an average of 1 year
  Tactile sensory evaluation was performed with Semmes-Weinstein Monofilaments.
Foot load distribution | Through study completion, an average of 1 year
  Diagnostic Support Baropodometer Footscan® 3D system will be used for static and dynamic pedobarographic analysis.
Balance | Through study completion, an average of 1 year
  Biodex Balance System will be used for static balance assessment. Functional reach test will be used for dynamic balance assessment. The child will be asked to stand sideways against the wall. Marking will be made from the tip of the third finger, with the child's arm flexed at 90 degrees. The child will be asked to reach forward as far as he can without taking a step, lifting his heels off the ground, and without changing his arm position. The third fingertip will be marked again and the distance between the two marks will be measured in centimeters

SECONDARY OUTCOMES:
Foot posture | Through study completion, an average of 1 year
  Foot posture analysis will be evaluated using the Foot Posture Index.
Quality of life assessment | Through study completion, an average of 1 year
  Children's quality of life will be evaluated with the 'Pediatric Quality of Life Inventory'.This scale is a quality of life scale that evaluates children's physical and psychosocial experiences. Turkish validity and reliability studies have been conducted.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided